CLINICAL TRIAL: NCT02163460
Title: Comparative Study Between the Use of Tubular Drains in Closed Suction System and the Use of Progressive Tension Sutures in Prevention of Infection and Seromas After Surgical Repair of Large Incisional Hernias
Brief Title: Repair of Large Incisional Hernias - To Drain or Not to Drain Randomised Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Estadual do Oeste do Paraná (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 009/2011-CEP
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Ventral Hernia
Keywords: ventral hernia; seroma; drainage; infection
MeSH Terms: conditions — Hernia, Ventral; Seroma; Infections | interventions — Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drain (Experimental): In group 1(Drain), a 4.8 mm diameter continuous closed-suction tubular drain : was placed between the aponeurosis and the subcutaneous tissue caudally to the incision.
  Interventions: Procedure: Drain
- Progressive Tension Sutures (Experimental): Drains were not used in group 2, but separate absorbable polyglactin 920 2/0 sutures were placed from the subcutaneous mesh to the aponeurosis every 2 cm by means of the progressive tension suture (or Quilting Sutures) technique, as described by Pollock et al
  Interventions: Procedure: Progressive Tension Sutures

INTERVENTIONS:
Procedure: Drain — In group 1, a 4.8 mm diameter continuous closed-suction tubular drain (Medsharp Ind.Com.Prod.Hosp.Ltda - reg. MS (Ministério da Saúde [Health Ministry registry]): 80267170001) was placed between the aponeurosis and the subcutaneous tissue caudally to the incision.
  Other Names: 4.8 mm diameter surgical closed-suction tubular drain
  Arms: Drain
Procedure: Progressive Tension Sutures — Drains were not used in group 2, but separate absorbable polyglactin 920 2/0 sutures were placed from the subcutaneous mesh to the aponeurosis every 2 cm by means of the progressive tension suture (or Quilting Sutures) technique, as described by Pollock et al
  Other Names: Quilting Sutures, Baroudi Sutures
  Arms: Progressive Tension Sutures

SUMMARY:
The aim of this study was to perform a randomised clinical trial comparing the use of closed-suction tubular drains and progressive tension sutures in individuals with large incisional hernias subjected to onlay mesh repair to evaluate the occurrence of seroma and surgical wound infection after surgery.

DETAILED DESCRIPTION:
The present randomised clinical trial was approved by the research ethics committees of the São Paulo School of Medicine - Federal University of São Paulo (Universidade Federal de São Paulo - UNIFESP), the State University of Western Paraná (Universidade Estadual do Oeste do Paraná - UNIOESTE) and the University Hospital of Western Paraná (Hospital Universitário do Oeste do Paraná - HUOP) in compliance with the 1964 Declaration of Helsinki and later updates.

The study design and randomisation followed the Consolidated Standards of Reporting Trials (CONSORT) version 2010 15.

All the participants read and signed an informed consent form at the preoperative assessment visit.

Inclusion and exclusion criteria Individuals with primary or recurrent incisional hernia were assessed at HUOP, and those with longitudinal or transverse ventral hernia secondary to a previous surgical incision, measuring 5 to 15 cm after dissection of the hernial sac and classified as large or very large according to Chevrel's classification, were considered to be eligible16. In individuals with multiple defects, the length between the cranial margin of the most cranial defect and the caudal margin of the most caudal defect was considered17. Individuals subjected to emergency surgery, with infection, immunosuppressed, younger than 18 or older than 80 years old, ASA III or IV, with a serum albumin concentration lower than 3.0 g/dl or who refused participation were excluded from the study.

Surgical technique The participants were admitted to the hospital the night before surgery to perform or update the assessment of their surgical risk according to the American Society of Anesthesiologists (ASA) criteria, as well as for measurement of the serum albumin concentration.

Incisional herniorrhaphy surgery was performed following the group's technique systematisation by a resident physician supervised by one of four surgeons professors at the medical course of UNIOESTE and who the using the onlay technique as described by Chevrel18-20. Antibiotic prophylaxis was performed with a single 2 g dose of cefazolin at the time of anaesthetic induction followed by a booster 1 g dose when the surgery lasted more than three hours.

The aponeurosis was dissected 5 cm beyond the aponeurotic defect. Approximation of the aponeurotic margins for midline reconstruction was performed using polyglactin 910 #1 sutures. Tension was relieved by releasing incisions performed on the external oblique muscle aponeurosis, 3 cm away from the linea alba, as described by Gibson21. A macroporous polypropylene monofilament P1 mesh of 100 g/m2 (Cousin Biotec) was fixed on the aponeurosis by separate 2-0 polypropylene sutures performed every 2 cm.

The participants were randomised immediately after mesh fixation by a computer-based random number generator and allocated to the two intervention groups.

Interventions In group 1, a 4.8 mm diameter continuous closed-suction tubular drain (Medsharp Ind.Com.Prod.Hosp.Ltda - reg. MS (Ministério da Saúde [Health Ministry registry]): 80267170001) was placed between the aponeurosis and the subcutaneous tissue caudally to the incision. Next, the subcutaneous tissue approximation was performed with separate absorbable polyglactin 910 2/0 sutures.

Drains were not used in group 2, but separate absorbable polyglactin 920 2/0 sutures were placed from the subcutaneous mesh to the aponeurosis every 2 cm by means of the progressive tension suture (or Quilting Sutures) technique, as described by Pollock et al.10-13.

Skin closure was performed with simple separate sutures at 1 cm intervals using nylon monofilament suture #4-0 in both groups. The participants were requested to use the support girdles provided by the surgical staff at the hospital and at home during the first 30 days after surgery.

In group 1, the drains were removed when the drained volume was less than 40 ml/24 hours.

Outcomes All the participants were clinically assessed by the attending staff to detect postoperative complications, seroma formation and surgical site infection, especially on postoperative (PO) days one, three, five, seven, 14-16 and 29-31. The data were recorded on a pre-established form.

All the participants were subjected to abdominal wall ultrasound to assess seroma formation at three time points defined as: early (PO days four to six), intermediate (PO days 14 to 16) and late (PO days 29 to 31). The tests were performed by the radiology staff at HUOP. Seroma was defined as the collection of any volume of subcutaneous fluid without debris. All the participants remained in the hospital until the first ultrasound assessment was performed. The presence of seroma was considered as the main outcome. Clinical seroma was defined as a visible bulge or fluctuation without signs of infection, subclinical seroma was defined as the absence of detectable abnormalities on physical examination but the presence of any volume of fluid collection on abdominal wall ultrasound, and seroma was defined as all occurrences of fluid collection detected on ultrasound.

Surgical wound infection was prospectively defined according to the criteria formulated by the Centers for Disease Control and Prevention (CDC) in the Guideline for Prevention of Surgical Site Infection, 1999 22.

Sample size calculation The sample size was calculated based on significance level alpha = 5% and 80% power. A two-tailed test for the comparison of the two proportions was used to compare the occurrence of seroma between the groups with drains (50.0%) or progressive tension sutures (10.0%)

Statistics The initial statistical analysis of all the data collected in the present study was descriptive. In regard to the quantitative (numerical) variables, summary measures including mean, standard deviation, median, maximum and minimum values were calculated, and one-dimensional scatterplots were constructed. The data corresponding to the qualitative (categorical) variables were assessed as absolute and relative (percent) frequencies.

Inferential analysis was performed to confirm or refute the evidence found in the descriptive analysis. For that purpose, Student's t-test for independent samples was used to compare the groups of participants.

In the inferential analysis, the significance level (α) was established as 5%. The statistical analyses were performed using software R version 2.15.2.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with primary or recurrent incisional hernia were assessed at HUOP, and those with longitudinal or transverse ventral hernia secondary to a previous surgical incision, measuring 5 to 15 cm after dissection of the hernial sac and classified as large or very large according to Chevrel's classification, were considered to be eligible.
* In individuals with multiple defects, the length between the cranial margin of the most cranial defect and the caudal margin of the most caudal defect was considered

Exclusion Criteria:

* Individuals subjected to emergency surgery, with infection
* Immunosuppressed
* Younger than 18 or older than 80 years old
* ASA III or IV, with a serum albumin concentration lower than 3.0 g/dl or who refused participation were excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Seroma | 1 month
  Clinical and/or radiological diagnosis of seroma until 1 month

SECONDARY OUTCOMES:
Infection | 1 month
  Surgical wound infection was prospectively defined according to the criteria formulated by the Centers for Disease Control and Prevention (CDC) in the Guideline for Prevention of Surgical Site Infection, 1999 in the first month postoperative

OTHER OUTCOMES:
hernia recurrence | 1 year
  clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Andre P Westphalen, MD, Principal Investigator — Universidade Estadual do Oeste do Paraná
Locations (1):
- Western Paraná State University / Universidade Estadual do Oeste do Paraná, Cascavel, Paraná, Brazil